CLINICAL TRIAL: NCT06418178
Title: A Dose Optimization Study of MDMA-Assisted Therapy for PTSD in U.S. Veterans
Brief Title: Dose Optimization of MDMA-Assisted Therapy for PTSD
Acronym: DosOp
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bronx VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rachel Yehuda, Mental Health Patient Care Center Director, Bronx VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 171633
Record Dates: First submitted 2024-05-06; First posted 2024-05-17 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; MDMA-Assisted Therapy; Dose Optimization; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Open label, within-subjects treatment arm. Participants receive 120mg + optional 60mg supplement. There will be from one to five dosing sessions that occur three to five weeks apart. Each dosing session is followed by three integration psychotherapy sessions.
  Interventions: Drug: Midomafetamine; Behavioral: Psychotherapy

INTERVENTIONS:
Drug: Midomafetamine — One to five MDMA-assisted therapy sessions, each followed by three non-drug psychotherapy sessions (see behavioral intervention below)
  Other Names: MDMA; 3,4-methylenedioxymethamphetamine
Behavioral: Psychotherapy — Standardized psychotherapy performed by therapy team

SUMMARY:
This open label, within-subjects dose optimization trial will investigate the optimal number of MDMA-Assisted Therapy treatment cycles (i.e., one MDMA session and three integration sessions) in a sample of U.S. veterans with PTSD. Participants will complete from one to five cycles of MDMA-AT.

DETAILED DESCRIPTION:
This open label, within-subjects dose optimization study will determine the optimal number of treatment cycles of MDMA-AT (one cycle consists of one Experimental Session followed by three Integrative Sessions) for significant improvement in a sample of U.S. veterans with PTSD. All participants will receive three non-drug preparatory sessions and at least one cycle of MDMA-assisted therapy with a team of two therapists. Each cycle will consist of one approximately 8-hour drug session followed by three 90-minute non-drug integrative sessions. After each cycle, participants will determine, in consultation with their therapy team, whether to continue with an additional cycle or to discontinue treatment. The decision will reflect the participant's perception of the potential for continued improvement (e.g., as based on current symptom burden, treatment response to date) weighed against the burden of an additional cycle (e.g., time required, any adverse events or emotional burden). Participants may complete up to a maximum of five cycles. The dose optimizing design allows for the identification of the optimal number of MDMA-AT cycles to achieve the best response and to assess tolerability of multiple cycles of MDMA-AT. Participants will also provide blood samples to be banked for future analysis of biological markers associated with treatment response.

For each participant, the study will consist of:

* Screening Period: initial screen, informed consent, eligibility assessment
* Enrollment Period with Enrollment Confirmation: Enrollment and medication tapering period (if needed) followed by psychological assessment and Enrollment Confirmation, collection of biomarker blood samples.
* Treatment Period: 3 Preparatory sessions; one to five Experimental Sessions, each followed by 3 non-drug Integrative Sessions and a follow-up visit with study therapists
* Post-treatment Period and Study Termination: Psychological Evaluation, biomarker blood samples, study termination visit

ELIGIBILITY:
Inclusion Criteria:

1. Are a U.S. military veteran at least 18 years old.
2. Are able to provide written, informed consent.
3. Are able to swallow pills.
4. Agree to have study visits recorded, including Experimental Sessions, psychological assessments, and non-drug therapy sessions.
5. Must provide a contact who is willing and able to be reached by the investigators in the event of a participant becoming unwell or unreachable.
6. If able to become pregnant, must have a negative pregnancy test at study entry and prior to each Experimental Session, and must agree to use adequate contraceptive methods.
7. Must have a current PTSD diagnosis at screening and baseline.
8. Must not participate in any other interventional clinical trials for the duration of the study.
9. Must commit to medication dosing, therapy, and all study procedures.

Exclusion Criteria:

1. Are not able to give adequate informed consent.
2. Have a history of any medical condition, or any significant clinical finding on screening tests, that could make receiving a sympathomimetic drug harmful.
3. Have uncontrolled hypertension.
4. Have evidence or history of significant medical or psychiatric disorders.
5. Have symptomatic liver disease.
6. Have history of hyponatremia or hyperthermia.
7. Weigh less than 48 kilograms (kg).
8. Unable or unwilling to safely taper off prohibited psychiatric medication.
9. Abusing illegal drugs or alcohol.
10. Have received Electroconvulsive Therapy (ECT) or ketamine therapy within 12 weeks of enrollment.
11. Are pregnant or nursing or are able to become pregnant and are not practicing an effective means of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | From Baseline to Outcome Site Visit (up to ~27 weeks for participants who complete all five treatment cycles)
  The PCL-5 is a 20-item self-report questionnaire in which respondents indicate the presence and severity of PTSD symptoms per DSM-5. Participants indicate how much distress they have experienced due to each symptom on a five-point Likert-type scale (1=Not at all to 5=Extremely).

SECONDARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | From Pre-treatment Psychological Evaluation to Post-treatment Psychological Evaluation (up to ~28 weeks for participants who complete all five treatment cycles)
  The last month CAPS-5 is a semi-structured interview that assesses index history of DSM-5-defined traumatic event exposure and past-month symptom severity to produce a diagnostic score (presence vs. absence) and a PTSD Total Severity score. The CAPS-5 rates intrusion symptoms (intrusive thoughts or memories), avoidance, cognitive and mood symptoms, arousal and reactivity symptoms, duration and degree of distress and dissociation.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Yehuda, PhD, Principal Investigator — James J. Peters VA Medical Center; Amy Lehrner, PhD, Principal Investigator — James J. Peters VA Medical Center
Locations (1):
- James J. Peters VA Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No